CLINICAL TRIAL: NCT00327964
Title: Utility of Rapid Diagnostic Tests (RDTs) for Malaria in Kampala, Uganda
Brief Title: Rapid Diagnostic Tests (RDTs) for Malaria in Kampala, Uganda
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: NIH/DMID 05-0110
Record Dates: First submitted 2006-05-18; First posted 2006-05-19 (Estimated); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Febrile Illness; Malaria
Keywords: malaria; fever; Uganda; children; rapid diagnostic tests; RDTs; Africa
MeSH Terms: conditions — Malaria; Fever

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Dried blood spots on filter paper
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- study population: 601 children enrolled in an on-going longitudinal antimalarial treatment efficacy trial in Kampala, Uganda.

SUMMARY:
Malaria remains a disease that causes much death and sickness, especially in sub-Saharan Africa. An accurate, simple, and inexpensive method of diagnosing malaria is urgently needed. The purpose of this study is to evaluate a different diagnostic method compared to those most frequently used. The study may also identify the factors causing false positive and false negative results using the alternative method. Participants will be 600 Ugandan children aged 1-10 years who are enrolled in protocol 04-068. Those who develop a fever over the 12 month duration of the study will be tested for malaria by both the standard and the new methods. These tests will require a few drops of blood to be collected by finger prick. Subjects will be treated on the basis of standard diagnostic testing (i.e. expert microscopy).

DETAILED DESCRIPTION:
Malaria remains one of the most devastating infectious diseases, causing high morbidity and mortality especially in sub-Saharan Africa. The need for an accurate, simple, and inexpensive method to diagnose malaria has become increasingly urgent. Rapid diagnostic tests (RDTs), based on detection of Plasmodium antigens, may represent a more practical diagnostic tool than traditional light microscopy. This longitudinal study's objectives are (1) to evaluate the clinical performance (sensitivity, specificity, positive and negative predictive values) of RDTs, as compared with presumptive diagnosis and microscopy, for the diagnosis of malaria in children in Kampala, Uganda, and (2) to identify host and test factors that lead to false positive and false negative RDT results by comparison with polymerase chain reaction (PCR) analysis. Study subjects in this RDT study will have already been enrolled in a larger on-going longitudinal study of antimalarial drug efficacy, tolerability, and safety that began at the Kampala study site in late 2004. In the RDT study, over a one-year period, study participants' blood samples will be evaluated with the current gold standard for malaria diagnosis (microscopy) as well as two types of RDT whenever they present with a new fever episode (the first fever after study enrollment, or a fever that occurs more than 14 days after the patient's most recently diagnosed episode of malaria). As part of the on-going longitudinal drug efficacy trial, probability sampling was used to select a random sample of 600 children, who will be followed for three years for all their health-care needs. The RDT study will involve evaluation of the cohort over 12 months, beginning in approximately the third quarter of 2005. This protocol is a substudy of 04-068.

ELIGIBILITY:
Inclusion Criteria: Member of the cohort participating in clinical trial of antimalarial drug efficacy in Kampala, which was enrolled based on criteria including the following characteristics:

1. Ages 1-10 (at time of original enrollment)
2. Parents' or guardians' agreement to bring the child to the study clinic for any fevers or other illnesses
3. Agreement to avoid medications administered outside the study
4. Intention to remain in Kampala for the full study period
5. Native Ugandan

Exclusion Criteria:

1. Presence of any known serious chronic disease (e.g. AIDS, sickle cell disease, malignancy)
2. Serious side effects to study medications used in cohort clinical trial of antimalarial drug efficacy

Ages: 1 Year to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 601 children enrolled in a longitudinal antimalarial treatment efficacy trial in Kampala, Uganda.
Sampling Method: Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2005-10; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
RDT accuracy

CONTACTS AND LOCATIONS:
Overall Officials: Heidi Hopkins, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- Mulago Hospital, Kampala, Uganda

REFERENCES:
- [Result] Hopkins H, Kambale W, Kamya MR, Staedke SG, Dorsey G, Rosenthal PJ. Comparison of HRP2- and pLDH-based rapid diagnostic tests for malaria with longitudinal follow-up in Kampala, Uganda. Am J Trop Med Hyg. 2007 Jun;76(6):1092-7. PMID 17556616
- See also: research collaboration website — http://www.muucsf.org